CLINICAL TRIAL: NCT01490203
Title: Pre-Surgical Treatment or Radio Frequency Ablation (RFA) Evaluation of Future Remnant Liver Function Using Gd-EOB-DTPA Enhanced MRI in Patients Undergoing Hepatic Resection /RFA for Hepatocellular Carcinoma
Brief Title: Evaluation of Remnant Liver Function Using Primovist-enhanced MRI Before Resection/Ablation of Hepatocellular Carcinoma
Acronym: LiFE
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bayer (Industry); Seoul St. Mary's Hospital (Other); Asan Medical Center (Other); Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Associate Professor, Seoul National University Hospital
Other Study IDs: LIFE_ISS_2011
Record Dates: First submitted 2011-12-07; First posted 2011-12-12 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Hepatocellular; Liver Dysfunction
Keywords: Gd-EOB-DTPA; MRI; Hepatectomy; Hepatocellular Carcinoma; Liver Function Tests
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: HCC resection/RFA: Patients who will undergo resection of at least two hepatic segments for HCC or radiofrequency ablation (RFA) for HCC and underwent gadoxetic acid (Gd-EOB-DTPA)-enhanced MRI
  Interventions: Drug: Gd-EOB-DTPA; Procedure: MRI
- Group 2: Potential liver donor: Potential liver donors with normal hepatic function and and underwent gadoxetic acid (Gd-EOB-DTPA)-enhanced MRI
  Interventions: Drug: Gd-EOB-DTPA; Procedure: MRI

INTERVENTIONS:
Drug: Gd-EOB-DTPA — 1. Gd-EOB-DTPA enhanced MRI will be obtained within 1 week before, and within 3 to 5 days after surgical resection of the liver.
  2. Gd-EOB-DTPA will be administered intravenously with an amount of 0.1mL/kg, 1mL/sec injection rate, followed by saline infusion.
  Other Names: Gadoxetic Acid Disodium; Primovist/Eovist; BAY86-4873
  Groups: Group 1: HCC resection/RFA
Drug: Gd-EOB-DTPA — 1. Gd-EOB-DTPA enhanced MRI will be performed within 3 days of obtaining ICG R15 test.
  2. Gd-EOB-DTPA will be administered intravenously with an amount of 0.1mL/kg, 1mL/sec injection rate, followed by saline infusion.
  Other Names: Gadoxetic Acid Disodium; Primovist/Eovist; BAY86-4873
  Groups: Group 2: Potential liver donor
Procedure: MRI — 1. Gd-EOB-DTPA enhanced MRI will be obtained within 1 week before, and within 3 to 5 days after surgical resection of the liver.
  2. Multiphasic MRI including dynamic hepatocyte specific phase will be performed for evaluation of hepatic extraction fraction, with 25 phase dynamic MRI obtained until 30 minutes after contrast injection.
  Groups: Group 1: HCC resection/RFA
Procedure: MRI — 1. Gd-EOB-DTPA enhanced MRI will be performed within 3 days of obtaining ICG R15 test.
  2. Multiphasic MRI including dynamic hepatocyte specific phase will be performed for evaluation of hepatic extraction fraction, with 25 phase dynamic MRI obtained until 30 minutes after contrast injection.
  Groups: Group 2: Potential liver donor

SUMMARY:
The purpose of this study is to determine whether the global and segmental hepatic uptake and excretion of Gd-EOB-DTPA on Gd-EOB-DTPA-enhanced liver MRI correlates with standard liver function test results in the patients with Hepatocellular Carcinoma (HCC) before major hepatic resection or radiofrequency ablation (RFA).

DETAILED DESCRIPTION:
1. Preoperative/RFA assessment of remnant liver function is important for avoiding posthepatectomy liver failure. However, the function of the future remnant is decreased in patients with chronic liver disease or cirrhosis, compared to that of healthy patients with an equal volume. Therefore, volume-based estimation of hepatic reserve function is inadequate for patients with hepatic dysfunction.
2. Standard clinical liver function tests, such as ICG clearance rate or Child-Pugh score, provides measurements of the global hepatic function, but cannot evaluate the functional distribution in the liver. Gd-EOB-DTPA (Gadoxetic acid, Primovist®, Bayer Schering) enhanced MRI has been recently demonstrated to have the potential to be an imaging-based liver function test, with the possibility to detect functional differences on a regional or even segmental level.
3. Gd-EOB-DTPA-enhanced liver MRI may be able to assess not only global but also segmental liver function in patients with hepatocellular carcinoma (HCC) who have a relatively high risk for developing liver failure after surgical resection due to coexistent hepatic damage by chronic viral hepatitis and/or cirrhosis preoperatively.

The purpose of this study is to determine whether the global and segmental hepatic uptake and excretion of Gd-EOB-DTPA on Gd-EOB-DTPA-enhanced liver MRI correlates with standard liver function test results in the patients with HCC before major hepatic resection/RFA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of HCC based on noninvasive diagnostic criteria of HCC proposed by 2010 AASLD
2. Surgical resection of hepatic resection greater than 2 Couinaud segments (including total hepatectomy for transplantation) or radiofrequency ablation is planned
3. Patients who provided the informed consent

Exclusion Criteria:

1. Patients younger than 18 yrs old
2. Patients who received hepatic surgery prior to this study
3. Patients who underwent TACE or RFA for greater than 2 segments within 3 months prior to this study
4. Patients who received radiation treatment including the liver or systemic chemotherapy
5. Patients who underwent contrast enhanced liver MRI within 3 days prior to this study
6. Patients with severe renal dysfunction (Cr .2.5 mg/dL or GFR < 30mL/min)
7. Patients with hypersensitivity to gadolinium
8. Patients with uncorrectable hypokalemia
9. Pregnant women, or reproductive age women who will not agree with contraception during this study period.
10. Patients with mental disorder which will interfere with voluntary agreement
11. Patients who have any contraindication to MRI (cardiac pacemaker, ferromagnetic implants, etc.)
12. Any other condition which, in the opinion of the Investigator, would make the patient unsuitable for enrollment or could interfere with the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients who will undergo hepatic resection/RFA for HCC. Group 2: Potential liver donors with normal hepatic function.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Correlation of hepatic extraction fraction (HEF) of future remnant liver function (RLF) obtained from Gd-EOB-DTPA enhanced MRI with postoperative ICG R15 clearance test results | 3 days (upto 5 days) after surgery
  Predicted RLF (HEF mL) = the sum of the individual HEF of each voxel in future remnant segment

SECONDARY OUTCOMES:
Correlation of various functional and volumetric parameters derived from Gd-EOB-DTPA enhanced MRI and clinical liver function tests obtained before and after surgical resection | within 7 days before, and 3 to 5 days after surgery
  1. Functional parameters derived from Gd-EOB-DTPA enhanced MRI include hepatic extraction fraction [HEF], input-relative blood flow [irBF], hepatocellular uptake index [HUI], liver to spleen ratio (LSR).
  2. Volumetric parameters include global liver volume and remnant liver volume.
  3. Clinical liver function tests include ICG R15, MELD score and Child-Pugh score.
  4. ICG R15 [Indocyanine green retention at 15 minutes, %] test will be performed within 3 days of preoperative MRI and 3 days after surgical resection.
Analysis of clinical and MRI parameters of postoperative complication and morbidity | upto 3 months (plus minus 1 week) after discharge
  1. Clinical parameters refer to the following.
     * Frequency of POD#5 days 50-50 criteria
     * Evaluation of operation related complication
     * Incidence of hepatic failure or death
  2. Functional and volumetric MRI parameters of patients with postoperative complication and morbidity will be evaluated.
  3. Correlation of MRI parameters with laboratory liver function tests.
Exploratory analysis of MRI parameters and ICG R15 derived from potential liver donors | within 3 days of ICG R15 test
  1. Correlation of functional parameters derived from Gd-EOB-DTPA enhanced MRI with ICG R15
  2. Correlation of functional and volumetric parameters derived from Gd-EOB-DTPA enhanced MRI
  3. Correlation of volumetric parameters derived from Gd-EOB-DTPA enhanced MRI and ICG15
  4. Comparison of functional MRI parameters between potential liver donors and patients undergoing hepatic resection for HCC.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Cheonnam University Hwasun Hospital, Hwasun-Gun, Cheonnam Province
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon JH, Choi JI, Jeong YY, Schenk A, Chen L, Laue H, Kim SY, Lee JM. Pre-treatment estimation of future remnant liver function using gadoxetic acid MRI in patients with HCC. J Hepatol. 2016 Dec;65(6):1155-1162. doi: 10.1016/j.jhep.2016.07.024. Epub 2016 Jul 28. PMID 27476767